CLINICAL TRIAL: NCT04276467
Title: Development and Validation of the International Classification of Functioning Disability and Health (ICF) Based Amputee Mobility Scale
Brief Title: Development of the ICF Based Amputee Mobility Scale
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Yasin Ekinci, MSc, Hacettepe University
Other Study IDs: GO 19/773
Record Dates: First submitted 2020-02-18; First posted 2020-02-19 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Amputation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lower limb amputation is a condition that reduces individuals' independence in daily life. Therefore, the main purpose of the rehabilitation process is to reintegrate the person as an independent and productive person as soon as possible. Although scales are frequently used in mobility evaluation in the clinic, they do not measure the advanced activities of patients. Therefore, the aim of the study is to obtain a comprehensive scale evaluating mobility in amputee. The mobility scale will be created using the two-round Delphi method. ICF (International Classification of Functioning Disability and Health) created by the World Health Organization, mobility subheading will be evaluated, and the questions that will be included in the scale will be compiled. In line with the data to be obtained from experts, a scale will be created.Scale and gold standard tests will be applied to patients so that validation of the scale will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral and traumatic lower limb loss
* Prosthesis use for at least 6 months

Exclusion Criteria:

* Not speaking or understanding Turkish
* Not having cognitive skills to perform the tests

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Lower Limb Amputee
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
2 Minute Walk Test | 3 March 2021
Amputee Mobility Predictor | 3 March 2021